CLINICAL TRIAL: NCT02323880
Title: A Phase 1 Study of Selinexor (KPT-330), A Selective XPO1 Inhibitor, in Recurrent and Refractory Pediatric Solid Tumors, Including CNS Tumors
Brief Title: Selinexor in Treating Younger Patients With Recurrent or Refractory Solid Tumors or High-Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1414; NCI-2014-02410 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1414; ADVL1414 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1414 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2014-12-16; First posted 2014-12-24 (Estimated); Results first posted 2024-01-02 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Malignant Glioma; Recurrent Brain Neoplasm; Recurrent Childhood Central Nervous System Neoplasm; Recurrent Childhood Glioblastoma; Recurrent Lymphoma; Recurrent Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Primary Central Nervous System Neoplasm; WHO Grade 3 Glioma
MeSH Terms: conditions — Glioma; Brain Neoplasms; Central Nervous System Neoplasms; Astrocytoma; Lymphoma | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selinexor) (Experimental): Patients receive selinexor PO on either a twice weekly (days 1, 3, 8, 10, 15, 17) or once weekly (days 1, 8, 15, and 22) schedule. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Pharmacological Study; Drug: Selinexor

INTERVENTIONS:
Other: Pharmacological Study — Correlative studies
Drug: Selinexor — Given PO
  Other Names: ATG-010; CRM1 Nuclear Export Inhibitor KPT-330; KPT 330; KPT-330; KPT330; Nexpovio; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330; Xpovio

SUMMARY:
This phase I trial studies the side effects and best dose of selinexor in treating younger patients with solid tumors or central nervous system (CNS) tumors that have come back (recurrent) or do not respond to treatment (refractory). Drugs used in chemotherapy, such as selinexor, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) or the maximum tolerated dose (MTD) of the tablet formulation of selinexor in children with recurrent/refractory solid and CNS tumors.

II. To describe the toxicities of selinexor in children with recurrent/refractory solid and CNS tumors.

III. To characterize the pharmacokinetics of the tablet formulation of selinexor in children with recurrent/refractory solid and CNS tumors.

SECONDARY OBJECTIVES:

I. To determine the antitumor effect of selinexor in a preliminary manner in children with recurrent/refractory solid and CNS tumors.

II. To determine the pharmacodynamic properties of selinexor in children and adolescents with refractory solid tumors in plasma proteins and whole blood ribonucleic acid (RNA).

III. To explore the penetration, pharmacodynamic effects, and biologic effects of selinexor in tumor tissue of patients with recurrent/refractory high-grade gliomas (HGG) requiring resection.

IV. To further assess the toxicity and antitumor effects of selinexor in children with recurrent/refractory HGG in expanded cohorts following dose-escalation by measuring rate of objective radiographic response (medical patients) and rate of progression-free survival (PFS) six months from the start of treatment (surgical patients).

OUTLINE: This is a dose escalation study.

Patients receive selinexor orally (PO) on either a twice weekly (days 1, 3, 8, 10, 15, 17) or once weekly (days 1, 8, 15, and 22) schedule. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a body surface area (BSA) >= 0.84 m^2
* Diagnosis:

  * Part A: Patients with recurrent or refractory solid tumors, including lymphoma and CNS tumors, are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG)
  * Part B: Patients with recurrent or refractory high grade glioma (World Health Organization [WHO] grade III/IV) including disseminated tumors (excluding diffuse intrinsic pontine glioma [DIPG]), not requiring surgical resection; patients must have had histologic verification of malignancy at original diagnosis or relapse
  * Part C: Patients with recurrent or refractory high grade glioma (WHO grade III/IV) and requiring surgical resection (excluding DIPG and disseminated tumors), who in the opinion of treating physicians, are medically stable to receive 2 doses of selinexor (8-10 days of treatment) before undergoing surgery without compromising the success of the procedure; note that if, in the opinion of treating physicians, current symptoms necessitate surgery before 2 doses will be able to be received, surgery should not be delayed to administer selinexor, and the patient would be ineligible for protocol therapy
* Disease status:

  * Part A: Patients must have either measurable or evaluable disease
  * Parts B and C: Patients must have measurable disease on imaging
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * External beam radiation therapy (XRT): At least 14 days after local palliative XRT (small port); at least 150 days must have elapsed if prior total body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis; at least 42 days must have elapsed if other substantial bone marrow (BM) radiation
  * Stem cell infusion without TBI: No evidence of active graft vs. host disease and at least 56 days must have elapsed after transplant or stem cell infusion
  * Patients must not have received prior exposure to selinexor
* For patients with solid tumors without known bone marrow involvement:
* * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* * Hemoglobin >= 8.0 g/dL at baseline (may receive red blood cell [RBC] transfusions)
* Patients with known bone marrow metastatic disease will be eligible for study if they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity; at least 5 of every cohort of 6 patients must be evaluable for hematologic toxicity for the dose-escalation part of the study; if dose-limiting hematologic toxicity is observed, all subsequent patients enrolled on Part A must be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or
* A serum creatinine based on age/gender as follows:

  * =< 0.6 mg/dL (patients age 1 to < 2 years)
  * =< 0.8 mg/dL (patients age 2 to < 6 years)
  * =< 1 mg/dL (patients age 6 to < 10 years)
  * =< 1.2 mg/dL (patients age 10 to < 13 years)
  * =< 1.4 mg/dL (female patients age >= 13 years)
  * =< 1.5 mg/dL (male patients age 13 to < 16 years)
  * =< 1.7 mg/dL (male patients age >= 16 years)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN = 135 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* Serum amylase =< 1.5 x ULN
* Serum lipase =< 1.5 x ULN
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* Patients must be able to swallow tablets whole
* Part C: Archived paraffin-embedded tissue (20 unstained slides or a tumor block) from a prior resection must be available as a control for correlative studies; if tissue blocks or slides are unavailable, the study chair must be notified prior to enrollment
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study, since there is yet no available information regarding human fetal or teratogenic toxicities; based on its mechanism of action and findings in animals, selinexor may cause fetal harm when administered to a pregnant woman; pregnancy tests must be obtained in girls who are post-menarchal; males with female partners of reproductive potential or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control- including a medically accepted barrier method of contraceptive method (e.g., male or female condom) for the entire period in which they are receiving protocol therapy and for at least 1 week following their last dose of study drug; abstinence is an acceptable method of birth control
* Concomitant medications

  * Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Investigational drugs: Patients who are currently receiving another investigational drug are not eligible
  * Anti-cancer agents: Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients with body mass index (BMI) < 3rd percentile for age, as defined by WHO criteria for patients 1-2 years of age and Centers for Disease Control and Prevention (CDC) criteria for patients > 2 years of age, are not eligible
* Patients with grade 3 ataxia or grade >1 extrapyramidal movement disorder are not eligible
* Patients with known macular degeneration, uncontrolled glaucoma, or cataracts are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Glade-Bender, Principal Investigator — COG Phase I Consortium
Locations (23):
- United States (23):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Green AL, Minard CG, Liu X, Safgren SL, Pinkney K, Harris L, Link G, DeSisto J, Voss S, Nelson MD, Reid JM, Fox E, Weigel BJ, Glade Bender J. Phase I Trial of Selinexor in Pediatric Recurrent/Refractory Solid and CNS Tumors (ADVL1414): A Children's Oncology Group Phase I Consortium Trial. Clin Cancer Res. 2025 May 1;31(9):1587-1595. doi: 10.1158/1078-0432.CCR-24-2754. PMID 39998852

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Dose Level 1: 35 mg/m^2 of Selinexor PO twice weekly on a days 1 and 3 schedule (Mon/Wed, Tues/Thurs, or Wed/Fri) of a 28 day, or 8 dose course (Pre-amendment #1)
- Part A: Dose Level 1 (DL 1): 35 mg/m^2 of Selinexor PO twice weekly on a days 1 and 3 schedule (Mon/Wed, Tues/Thurs, or Wed/Fri) on Weeks 1-3, Week 4 rest, on a 28 day course (Amendment 1)
- Part A: Dose Level -1 (DL -1): 20 mg/m^2 of Selinexor PO twice weekly on a days 1 and 3 schedule (Mon/Wed, Tues/Thurs, or Wed/Fri) on Weeks 1-3, Week 4 rest, on a 28 day course
- Part A: Weekly Dose Level 1 (WDL 1): 45 mg/m^2 Selinexor once weekly, on days 1, 8, 15, and 22 of a 28-day cycle
- Part A: Weekly Dose Level -1 (WDL -1): 35 mg/m2 Selinexor once weekly, on days 1, 8, 15, and 22 of a 28-day cycle
- Part B: Weekly Dose Level -1 (WDL -1); Part PK: Weekly Dose Level -1 (WDL -1): 35 mg/m^2 Selinexor once weekly, on days 1, 8, 15, and 22 of a 28-day cycle
- Part PK: Dose Level -1 (DL -1): 20 mg/m2 of Selinexor PO twice weekly on a days 1 and 3 schedule (Mon/Wed, Tues/Thurs, or Wed/Fri) on Weeks 1-3, Week 4 rest, on a 28 day course
Period: Overall Study
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 1 (DL 1) | Part A: Dose Level -1 (DL -1) | Part A: Weekly Dose Level 1 (WDL 1) | Part A: Weekly Dose Level -1 (WDL -1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Dose Level -1 (DL -1) | Part PK: Weekly Dose Level -1 (WDL -1)
Started | 6 | 13 | 6 | 6 | 6 | 10 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 13 | 6 | 6 | 6 | 10 | 6 | 6
Not completed — Adverse Event | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 4 | 11 | 5 | 5 | 4 | 8 | 4 | 6
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: Dose Level 1 (DL1): 35 mg/m^2 of Selinexor PO twice weekly on a days 1 and 3 schedule (Mon/Wed, Tues/Thurs, or Wed/Fri) on Weeks 1-3, Week 4 rest, on a 28 day course (Amendment 1)
- Total: Total of all reporting groups
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 1 (DL1) | Part A: Dose Level -1 (DL -1) | Part A: Weekly Dose Level 1 (WDL 1) | Part A: Weekly Dose Level -1 (WDL -1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Dose Level -1 (DL -1) | Part PK: Weekly Dose Level -1 (WDL -1) | Total
Number analyzed (Participants) | 6 | 13 | 6 | 6 | 6 | 10 | 6 | 6 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 13 | 6 | 4 | 5 | 9 | 5 | 6 | 54
  Between 18 and 65 years | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 5
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 13.5 [11.0 to 18.0] | 16 [10.0 to 18.0] | 15.5 [6.0 to 17.0] | 16.5 [7.0 to 20.0] | 14 [7.0 to 20.0] | 15.5 [7.0 to 19.0] | 10.5 [7.0 to 20.0] | 11 [6.0 to 14.0] | 15 [6.0 to 20.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 3 | 4 | 5 | 3 | 3 | 4 | 33
  Male | 4 | 4 | 3 | 2 | 1 | 7 | 3 | 2 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 8
  Not Hispanic or Latino | 4 | 10 | 6 | 4 | 4 | 8 | 6 | 5 | 47
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 0 | 0 | 1 | 3 | 1 | 8
  White | 4 | 8 | 5 | 4 | 3 | 5 | 3 | 3 | 35
  More than one race | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 2 | 0 | 1 | 2 | 1 | 0 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities of Selinexor
Description: The number of toxicity evaluable patients experiencing a dose limiting toxicity at least possibly attributable to selinexor by study part, schema, and dose level.
Time Frame: Up to 28 days
Population: Toxicity evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 1 (DL 1) | Part A: Dose Level -1 (DL -1) | Part A: Weekly Dose Level 1 (WDL 1) | Part A: Weekly Dose Level -1 (WDL -1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Dose Level -1 (DL -1) | Part PK: Weekly Dose Level -1 (WDL -1)
Number analyzed (Participants) | 6 | 12 | 6 | 6 | 6 | 7 | 6 | 6
Participants | 0 | 4 | 1 | 2 | 1 | 0 | 2 | 0

2. Primary Outcome: Number of Adverse Events of Selinexor
Description: The number of patients experiencing adverse events at least possibly attributable to selinexor by study part, schema, and dose level.
Time Frame: Up to 6 years 11 months
Population: Toxicity evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 1 (DL 1) | Part A: Dose Level -1 (DL -1) | Part A: Weekly Dose Level 1 (WDL 1) | Part A: Weekly Dose Level -1 (WDL -1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Dose Level -1 (DL -1) | Part PK: Weekly Dose Level -1 (WDL -1)
Number analyzed (Participants) | 6 | 12 | 6 | 6 | 6 | 7 | 6 | 6
Participants | 6 | 12 | 6 | 6 | 6 | 7 | 6 | 6

3. Primary Outcome: Area Under the Drug Concentration Curve of Selinexor
Description: The median (min, max) of the area under the drug concentration curve evaluated at 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post dose on day 1 for Selinexor by study part, schema, and dose level.
Time Frame: Up to 2 days
Population: All eligible patients
Measure: Median (Full Range); unit: h*ng/ml
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 1 (DL 1) | Part A: Dose Level -1 (DL -1) | Part A: Weekly Dose Level 1 (WDL 1) | Part A: Weekly Dose Level -1 (WDL -1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Dose Level -1 (DL -1) | Part PK: Weekly Dose Level -1 (WDL -1)
Number analyzed (Participants) | 6 | 13 | 6 | 6 | 6 | 10 | 6 | 6
h*ng/ml | 5030 [3807.3 to 8789.4] | 4656.8 [3660.5 to 7285.5] | 2602.4 [2355.9 to 4889.3] | 6173.2 [5401.1 to 9161.2] | 7135.9 [4718.0 to 8665.6] | 4666.9 [2154.7 to 10151.4] | 3132.8 [2028.5 to 3377.1] | 6505.5 [4739.7 to 8809.0]

4. Secondary Outcome: Antitumor Effect of Selinexor
Description: Number of patients with best response using RECIST 1.1 criteria of partial response (at least a 30% decrease in the sum of the diameters of target lesions) or complete response (disappearance of all target and non-target lesions and any pathological lymph nodes must have reduction in short axis to <10 mm).
Time Frame: Up to 6 years 11 months
Population: Responsive patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 1 (DL 1) | Part A: Dose Level -1 (DL -1) | Part A: Weekly Dose Level 1 (WDL 1) | Part A: Weekly Dose Level -1 (WDL -1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Dose Level -1 (DL -1) | Part PK: Weekly Dose Level -1 (WDL -1)
Number analyzed (Participants) | 6 | 13 | 6 | 6 | 6 | 10 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Pharmacodynamics of Selinexor
Description: Median (min,max) ratio of XPO1 mRNA expression after treatment to pre-treatment by study part, schema, and dose
Time Frame: Up to 28 days
Population: There were 0 (zero) patients from Part A: Dose Level 1 (Pre-amendment #1). Participation in the PD studies was optional. The subjects who had matched pre- and post-treatment blood samples were analyzed; not all the subjects had samples collected for PD analysis.
Measure: Median (Full Range); unit: Ratio of XPO1 mRNA expression
Arm/Group | Part A: Dose Level 1 (DL 1) | Part A: Dose Level -1 (DL -1) | Part A: Weekly Dose Level 1 (WDL 1) | Part A: Weekly Dose Level -1 (WDL -1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Dose Level -1 (DL -1) | Part PK: Weekly Dose Level -1 (WDL -1)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 4 | 1 | 2
Ratio of XPO1 mRNA expression | 7.1 [7.1 to 7.1] | 4 [3.5 to 4.5] | 5.5 [4.2 to 6.7] | 1.7 [0.2 to 3.2] | 4.6 [1.2 to 5.3] | 7.9 [7.9 to 7.9] | 5.4 [5.0 to 5.9]

6. Secondary Outcome: Pharmacodynamics of Selinexor in High-grade Glioma (HGG) Patients
Description: Median (min,max) ratio of XPO1 mRNA expression after treatment to pre-treatment by study part, schema, and dose
Time Frame: Up to 28 days
Population: high-grade glioma (HGG) patients with data available
Measure: Median (Full Range); unit: Ratio of XPO1 mRNA expression
Arm/Group | Part A: Weekly Dose Level 1 (WDL 1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Weekly Dose Level -1 (WDL -1)
Number analyzed (Participants) | 1 | 4 | 1
Ratio of XPO1 mRNA expression | 4.2 [4.2 to 4.2] | 4.6 [1.2 to 5.3] | 5.9 [5.9 to 5.9]

7. Secondary Outcome: Radiographic Response of Selinexor in High-grade Glioma (HGG) Patients
Description: Number of HGG patients with radiographic response by study part, schema, and dose level.
Time Frame: Up to 6 years 11 months
Population: high-grade glioma (HGG) patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 1 (DL 1) | Part A: Weekly Dose Level 1 (WDL 1) | Part A: Weekly Dose Level -1 (WDL -1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Weekly Dose Level -1 (WDL -1)
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 9 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Progression-free Survival of Selinexor in Surgical High-grade Glioma (HGG) Patients
Description: Number of surgical HGG patients with 6-month progression-free survival using the Response Evaluation Criteria in solid tumors criteria (RECIST v1.1) defining best response of progressive disease including at least 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study and no prior stable disease, partial response, or complete response.
Time Frame: Up to 6 months
Population: high-grade glioma (HGG) patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 1 (DL 1) | Part A: Dose Level -1 (DL -1) | Part A: Weekly Dose Level 1 (WDL 1) | Part A: Weekly Dose Level -1 (WDL -1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Dose Level -1 (DL -1) | Part PK: Weekly Dose Level -1 (WDL -1)
Number analyzed (Participants) | 3 | 3 | 0 | 2 | 2 | 9 | 0 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 7 years 8 months
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Groups:
- Part A: Dose Level 1 (DL1)(Amendment 1): Amendment 1- 35 mg/m^2 of Selinexor PO twice weekly on a days 1 and 3 schedule (Mon/Wed, Tues/Thurs, or Wed/Fri) on Weeks 1-3, Week 4 rest, on a 28 day course (amendment #1)
- Part A: Dose Level -1 (DL-1): 20 mg/m^2 of Selinexor PO twice weekly on a days 1 and 3 schedule (Mon/Wed, Tues/Thurs, or Wed/Fri) on Weeks 1-3, Week 4 rest, on a 28 day course
- Part PK: Weekly Dose Level -1 (DL -1): 35 mg/m^2 Selinexor once weekly, on days 1, 8, 15, and 22 of a 28-day cycle
Arm/Group | Part A: Dose Level 1 | Part A: Dose Level 1 (DL1)(Amendment 1) | Part A: Dose Level -1 (DL-1) | Part A: Weekly Dose Level 1 (WDL 1) | Part A: Weekly Dose Level -1 (WDL -1) | Part B: Weekly Dose Level -1 (WDL -1) | Part PK: Dose Level -1 (DL -1) | Part PK: Weekly Dose Level -1 (DL -1)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/13 | 0/6 | 0/6 | 0/6 | 2/10 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 5/13 | 3/6 | 2/6 | 3/6 | 3/10 | 0/6 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 13/13 | 6/6 | 6/6 | 6/6 | 10/10 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Dose Level 1 (N=6) | Part A: Dose Level 1 (DL1)(Amendment 1) (N=13) | Part A: Dose Level -1 (DL-1) (N=6) | Part A: Weekly Dose Level 1 (WDL 1) (N=6) | Part A: Weekly Dose Level -1 (WDL -1) (N=6) | Part B: Weekly Dose Level -1 (WDL -1) (N=10) | Part PK: Dose Level -1 (DL -1) (N=6) | Part PK: Weekly Dose Level -1 (DL -1) (N=6)
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Edema cerebral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Dose Level 1 (N=6) | Part A: Dose Level 1 (DL1)(Amendment 1) (N=13) | Part A: Dose Level -1 (DL-1) (N=6) | Part A: Weekly Dose Level 1 (WDL 1) (N=6) | Part A: Weekly Dose Level -1 (WDL -1) (N=6) | Part B: Weekly Dose Level -1 (WDL -1) (N=10) | Part PK: Dose Level -1 (DL -1) (N=6) | Part PK: Weekly Dose Level -1 (DL -1) (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 4 | 3 | 2 | 0
Abducens nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Accessory nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acoustic nerve disorder NOS (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 8 | 5 | 1 | 5 | 5 | 2 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 0 | 2 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2 | 2 | 3 | 1 | 1
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 11 | 3 | 4 | 3 | 6 | 3 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 7 | 5 | 4 | 4 | 5 | 4 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 6 | 5 | 1 | 3 | 4 | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 4 | 1 | 1 | 2 | 2 | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 2 | 3 | 1 | 1
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 1
Blurred vision (Eye disorders) | 2 | 4 | 1 | 0 | 4 | 2 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac disorders - Other, ASYMPTOMATIC LV DSYFUNCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Concentration impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 5 | 3 | 3 | 5 | 3 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 2 | 3 | 1 | 1 | 2
Creatinine increased (Investigations) | 1 | 3 | 0 | 1 | 1 | 3 | 2 | 0
Cushingoid (Endocrine disorders) | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Delusions (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 6 | 3 | 2 | 4 | 3 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 5 | 1 | 1 | 5 | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 4 | 0 | 0 | 1 | 1 | 1 | 0
Dysesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 3 | 3 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0
Ear and labyrinth disorders - Other, EAR PRESSURE (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear and labyrinth disorders - Other, PHONOPHOBIA (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Edema face (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2
Eye disorders - Other, DECREASED VISION AND LIGHT PERCEPTION (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, DECREASED VISUAL ACUITY (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, DISCONJUGATE GAZE (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, DOUBLE VISION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, Double vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye disorders - Other, FIELD DEFICIT (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, MILD OPTIC ATROPHY (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, PARINAUD'S SYNDROME (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, PERIORBITAL PAIN (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, PTOSIS (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, Ptosis of left eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye disorders - Other, R ESOTROPIA (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, RIGHT APD (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, RIGHT EXTROPIA (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, RIGHT EYE SWELLING/PTOSIS (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, VISION LOSS (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, VISUAL FIELD DEFICIT (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 1 | 1 | 0 | 2 | 3 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 4 | 0 | 0 | 0 | 3 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Fatigue (General disorders) | 6 | 10 | 5 | 3 | 5 | 10 | 5 | 4
Fecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 4 | 2 | 1 | 1 | 3 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0
Gastrointestinal disorders - Other, ABDOMINAL CRAMPING (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, BRIGHT RED BLOOD PER RECTUM/POSSIBLE INTERNAL FISSURE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, TOOTH SENSITIVITY (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, ABDOMINAL CRAMPING (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, COLD INTOLERANCE (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, NIGHT SWEATS (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, OSMOPHOBIA (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, POLYDIPSIA (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, RHINORRHEA (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, surgical site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 1 | 1 | 1 | 0 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 9 | 2 | 2 | 2 | 6 | 3 | 3
Hearing impaired (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1
Hemoglobin increased (Investigations) | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatobiliary disorders - Other, NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 7 | 0 | 2 | 3 | 3 | 1 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 0 | 2 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 1 | 1 | 5 | 0 | 2
Hypernatremia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 1
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 5 | 1 | 1 | 3 | 6 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 6 | 1 | 2 | 1 | 2 | 0 | 3
Hypoglossal nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 4 | 4 | 3 | 1 | 3 | 1 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 0 | 1 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 6 | 2 | 2 | 3 | 4 | 1 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 5 | 3 | 2 | 4 | 3 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
INR increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other, CLOSTRIDIUM DIFFICILE (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infections and infestations - Other, INFLUENZA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, PARAINFLUENZA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, STREP PHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other, salmonella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, PSEUDOMENINGOCELE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 3 | 0 | 2 | 2 | 2 | 0
Intracranial hemorrhage (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, BICARBONATE < LLN (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BICARBONATE DECREASED (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BICARBONATE LOW (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BICARBONATE SERUM LOW (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, DECREASE CO2 (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, DECREASED CO2 (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, Decreased creatinine (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, ELEVATED BUN (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED LDH (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED TSH (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, Elevated Chloride (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, Elevated chloride (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Investigations - Other, HYPOCHLOREMIA (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, INCREASED CHLORIDE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LOW BICARB (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LOW BICARBONATE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LOW CO2 (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LOW TESTOSTERON (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 7 | 4 | 3 | 4 | 10 | 2 | 4
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolism and nutrition disorders - Other, (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, BICARBONATES (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, Bicarbonate, low (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, DIABETES INSIPIDUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metabolism and nutrition disorders - Other, HYPERPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, INCREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Movements involuntary (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscle weakness left-sided (Nervous system disorders) | 0 | 3 | 0 | 0 | 2 | 2 | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0
Muscle weakness right-sided (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 1
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, Achiness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, LEFT KNEE TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, RIGHT ANKLE TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 10 | 6 | 5 | 5 | 8 | 3 | 6
Neck edema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Nervous system disorders - Other, ACUTE NEURO CHANGES (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, HYPERALGESIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, LEFT SIDED DECREASED SENSORY AND PROPIOCEPTION (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, PSUEDOBALBAR AFFECT (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 5 | 10 | 6 | 6 | 5 | 7 | 5 | 5
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0
Oculomotor nerve disorder (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 2 | 1 | 5 | 4 | 2
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Papilledema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 4 | 1 | 2 | 1 | 2 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 5 | 11 | 5 | 4 | 6 | 6 | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Premature menopause (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 2 | 3 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 1
Psychiatric disorders - Other, ADHD (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psychiatric disorders - Other, AUTISIM (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, EMOTIONAL (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, HX OF ADHD (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 3 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, TONSILLITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 4 | 1 | 1 | 0 | 1 | 2 | 0 | 3
Serum amylase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 4 | 3 | 1 | 3 | 1 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, INCISION, LEFT OCCIPITAL REGION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, INCISION, RIGHT PARIETAL REGION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, NAIL BRITTLENESS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, NEVI (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, PEELING SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, PLANTAR WART (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, SCARRING (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, abrasions- bilateral lower extremity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 1 | 0 | 1 | 1
Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Surgical and medical procedures - Other, CRANIOTOMY (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, Portacath placement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 1 | 1
Trochlear nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 10 | 4 | 4 | 4 | 6 | 4 | 6
Weight gain (Investigations) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Weight loss (Investigations) | 4 | 3 | 3 | 2 | 2 | 2 | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 6 | 12 | 6 | 6 | 5 | 8 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT02323880/Prot_SAP_000.pdf